CLINICAL TRIAL: NCT04848831
Title: Diagnosis of Invasive Pulmonary Aspergillosis (IPA) - Specific Testing in Bronchial Secretions Versus Bronchoalveolar Fluid in Patients With and Without COVID-19
Brief Title: Diagnosis of Invasive Pulmonary Aspergillosis, Specific Testing in Bronchial Secretions Versus Bronchoalveolar Fluid
Acronym: DipA2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: DipA2
Record Dates: First submitted 2021-02-07; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Invasive Pulmonary Aspergillosis
Keywords: IPA; Aspergillus; Galactomannan; Aspergillus PCR; Aspergillus LFA; Bronchoscopy
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this research project is to compare the results of Aspergillus specific test methods Aspergillus Galactomannan Enzyme Immunoassay (GM-EIA), Aspergillus polymerase chain reaction (PCR), Aspergillus Galactomannan Lateral Flow Assay (LFA) from different respiratory tract secretions. The bronchoalveolar lavage (BAL) fluid and bronchial secretions (NBL) are compared in the same examination for each patient.

DETAILED DESCRIPTION:
Invasive pulmonary Infection with Aspergillus species has emerged as one of the most common causes of infectious death in critically ill patients (38%-79%). The incidence of invasive pulmonary Aspergillosis (IPA) in intensive care units is still not sufficiently clear and ranges between 0.3 % and 19 %. In the last two decades, IPA has been documented as an emerging disease in ICU patients without classic risk factors. The establishment of new therapeutic options in oncology with small-molecule kinase inhibitors (SMKI) and CAR (chimeric antigen receptor) T cell therapy have also led to an increase in IPA. Furthermore, during the influenza epidemics since 2009 and during the SARS-CoV-2 pandemic, IPA was observed in COVID-19 patients without classic risk factors. The cultural detection of molds can take between several days and up to 2 weeks, as this is a slow growing fungus. An Aspergillus Galactomannan EIA (enzyme immunoassay), an Aspergillus PCR (polymerase chain reaction) examination of the respiratory tract material is already available after 4-24 hours. A test using Aspergillus Galactomannan LFA (lateral flow assay) or LFD (lateral flow device) even furthers reduces this interval to 45 minutes. These tests allow the attending physician to initiate a much faster antimycotic treatment. Up to now, the samples for these examinations have been routinely obtained from bronchoscopically obtained bronchoalveolar lavage fluids. In this bronchoalveolar lavage (BAL), body-warm saline solution (NaCl) is instilled into segmental ostia of the lung and immediately re-aspirated . However, there are first indications that examinations from bronchial secretions using deep suction without bronchoscopy achieve similar results to the examination of the BAL. The bronchoscopic diagnosis in COVID-19 patients is probably associated with an increased risk of infection for the examiner due to the aerosol formation during this examination. Two studies from the first wave of the SARS-CoV-2 pandemic have therefore used secretions from the bronchial system = non-bronchoscopic lavage (NBL) to diagnose IPA. This method appears to be reasonable save, appropriate and less risky, but has never been scientifically validated for aspergillus infections. It is not yet clear whether the Aspergillus Galactomannan EIA, the Aspergillus PCR test and the Aspergillus LFA test provide comparable or transmissible results in both lung compartments. A direct comparison of the test results of the bronchoalveolar lavage (BAL) and the bronchial secretion (NBL) have not been described in the literature.

Study Design:

Monocentric prospective exploratory (and in the course confirmatory) cohort study.

1. st pilot phase: Pilot study to test the feasibility and to gain information for the case number calculation of a subsequent larger prospective study.
2. nd study phase: The statistically calculated number of patients who undergo a bronchoscopy during their stay at the UKE and who are urgently suspected of having IPA or who are confirmed to have IPA will be examined for bronchial secretions (NBL) and BAL fluids.

ELIGIBILITY:
Inclusion Criteria:

1. Age: at least 18 years
2. Consent to prospective data collection.
3. Clinical need for bronchoscopic examination.

Exclusion Criteria:

Refusal of consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4) Suspicion of invasive pulmonary aspergillosis:
  (a) Clinical:
  * Neutropenia
  * Hematooncological disease
  * Allogeneic stem cell transplantation
  * Organ transplantation
  * SARS-CoV-2
  * Influenza
    b) Radiological:
  * Aspergillus typical findings on computed tomography.
    c) Microbiological:
  * Aspergillus positive findings from respiratory tract secretions (culture, galactomannan, PCR) or d) Confirmed invasive pulmonary aspergillosis.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Equivalence of quantitative results of Aspergillus galactomannan EIA examination from bronchial secretions (NBL) and BAL in one patient. | The observation period for each individual patient begins with bronchoscopic examination (day 0) and ends after 90 days (day 90).
  The Aspergillus antigen findings (galactomannan-EIA) quantitative show now deviation

SECONDARY OUTCOMES:
Number of matched results (within a study participant) of Aspergillus PCR examination from BAL and NBL. | The observation period for each individual patient begins with bronchoscopic examination (day 0) and ends after 90 days (day 90).
  One patients results are same, positive or negative in both lung compartments (BAL and NBL).
Number of matched results (within a study participant) of Aspergillus galactomannan LFA examination from BAL and NBL. | The observation period for each individual patient begins with bronchoscopic examination (day 0) and ends after 90 days (day 90).
  One patients results are same, positive or negative in both lung compartments (BAL and NBL).

CONTACTS AND LOCATIONS:
Overall Officials: Maria Schroeder, MD, Principal Investigator — University Medical Center Hamburg-Eppendorf, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taccone FS, Van den Abeele AM, Bulpa P, Misset B, Meersseman W, Cardoso T, Paiva JA, Blasco-Navalpotro M, De Laere E, Dimopoulos G, Rello J, Vogelaers D, Blot SI; AspICU Study Investigators. Epidemiology of invasive aspergillosis in critically ill patients: clinical presentation, underlying conditions, and outcomes. Crit Care. 2015 Jan 12;19(1):7. doi: 10.1186/s13054-014-0722-7. PMID 25928694
- [Background] Loughlin L, Hellyer TP, White PL, McAuley DF, Conway Morris A, Posso RB, Richardson MD, Denning DW, Simpson AJ, McMullan R. Pulmonary Aspergillosis in Patients with Suspected Ventilator-associated Pneumonia in UK ICUs. Am J Respir Crit Care Med. 2020 Oct 15;202(8):1125-1132. doi: 10.1164/rccm.202002-0355OC. PMID 32609533
- [Background] Meersseman W, Van Wijngaerden E. Invasive aspergillosis in the ICU: an emerging disease. Intensive Care Med. 2007 Oct;33(10):1679-81. doi: 10.1007/s00134-007-0792-y. Epub 2007 Jul 24. No abstract available. PMID 17646965
- [Background] Latge JP, Chamilos G. Aspergillus fumigatus and Aspergillosis in 2019. Clin Microbiol Rev. 2019 Nov 13;33(1):e00140-18. doi: 10.1128/CMR.00140-18. Print 2019 Dec 18. PMID 31722890
- [Background] Wauters J, Baar I, Meersseman P, Meersseman W, Dams K, De Paep R, Lagrou K, Wilmer A, Jorens P, Hermans G. Invasive pulmonary aspergillosis is a frequent complication of critically ill H1N1 patients: a retrospective study. Intensive Care Med. 2012 Nov;38(11):1761-8. doi: 10.1007/s00134-012-2673-2. Epub 2012 Aug 16. PMID 22895826
- [Background] Schauwvlieghe AFAD, Rijnders BJA, Philips N, Verwijs R, Vanderbeke L, Van Tienen C, Lagrou K, Verweij PE, Van de Veerdonk FL, Gommers D, Spronk P, Bergmans DCJJ, Hoedemaekers A, Andrinopoulou ER, van den Berg CHSB, Juffermans NP, Hodiamont CJ, Vonk AG, Depuydt P, Boelens J, Wauters J; Dutch-Belgian Mycosis study group. Invasive aspergillosis in patients admitted to the intensive care unit with severe influenza: a retrospective cohort study. Lancet Respir Med. 2018 Oct;6(10):782-792. doi: 10.1016/S2213-2600(18)30274-1. Epub 2018 Jul 31. PMID 30076119
- [Background] van Arkel ALE, Rijpstra TA, Belderbos HNA, van Wijngaarden P, Verweij PE, Bentvelsen RG. COVID-19-associated Pulmonary Aspergillosis. Am J Respir Crit Care Med. 2020 Jul 1;202(1):132-135. doi: 10.1164/rccm.202004-1038LE. No abstract available. PMID 32396381
- [Background] Rutsaert L, Steinfort N, Van Hunsel T, Bomans P, Naesens R, Mertes H, Dits H, Van Regenmortel N. COVID-19-associated invasive pulmonary aspergillosis. Ann Intensive Care. 2020 Jun 1;10(1):71. doi: 10.1186/s13613-020-00686-4. No abstract available. PMID 32488446
- [Background] Nasir N, Farooqi J, Mahmood SF, Jabeen K. COVID-19-associated pulmonary aspergillosis (CAPA) in patients admitted with severe COVID-19 pneumonia: An observational study from Pakistan. Mycoses. 2020 Aug;63(8):766-770. doi: 10.1111/myc.13135. Epub 2020 Jul 18. PMID 32585069
- [Background] Koehler P, Cornely OA, Bottiger BW, Dusse F, Eichenauer DA, Fuchs F, Hallek M, Jung N, Klein F, Persigehl T, Rybniker J, Kochanek M, Boll B, Shimabukuro-Vornhagen A. COVID-19 associated pulmonary aspergillosis. Mycoses. 2020 Jun;63(6):528-534. doi: 10.1111/myc.13096. Epub 2020 May 15. PMID 32339350
- [Background] Dalhoff K, Abele-Horn M, Andreas S, Deja M, Ewig S, Gastmeier P, Gatermann S, Gerlach H, Grabein B, Heussel CP, Hoffken G, Kolditz M, Kramme E, Kuhl H, Lange C, Mayer K, Nachtigall I, Panning M, Pletz M, Rath PM, Rohde G, Rosseau S, Schaaf B, Schreiter D, Schutte H, Seifert H, Spies C, Welte T; Unter Mitwirkung der folgenden Wissenschaftlichen Fachgesellschaften und Institutionen: Deutsche Gesellschaft fur Chirurgie; Deutsche Gesellschaft fur Innere Medizin e. V.; Deutsche Gesellschaft fur Internistische Intensivmedizin und Notfallmedizin; Deutsche Sepsis-Gesellschaft e. V.; und Robert Koch-Institut. [Epidemiology, Diagnosis and Treatment of Adult Patients with Nosocomial Pneumonia - Update 2017 - S3 Guideline of the German Society for Anaesthesiology and Intensive Care Medicine, the German Society for Infectious Diseases, the German Society for Hygiene and Microbiology, the German Respiratory Society and the Paul-Ehrlich-Society for Chemotherapy, the German Radiological Society and the Society for Virology]. Pneumologie. 2018 Jan;72(1):15-63. doi: 10.1055/s-0043-121734. Epub 2018 Jan 16. German. PMID 29341032
- [Background] Lass-Florl C, Lo Cascio G, Nucci M, Camargo Dos Santos M, Colombo AL, Vossen M, Willinger B. Respiratory specimens and the diagnostic accuracy of Aspergillus lateral flow assays (LFA-IMMY): real-life data from a multicentre study. Clin Microbiol Infect. 2019 Dec;25(12):1563.e1-1563.e3. doi: 10.1016/j.cmi.2019.08.009. Epub 2019 Aug 22. PMID 31445208
- [Background] Van Biesen S, Kwa D, Bosman RJ, Juffermans NP. Detection of Invasive Pulmonary Aspergillosis in COVID-19 with Nondirected BAL. Am J Respir Crit Care Med. 2020 Oct 15;202(8):1171-1173. doi: 10.1164/rccm.202005-2018LE. No abstract available. PMID 32668167
- [Background] White PL, Dhillon R, Cordey A, Hughes H, Faggian F, Soni S, Pandey M, Whitaker H, May A, Morgan M, Wise MP, Healy B, Blyth I, Price JS, Vale L, Posso R, Kronda J, Blackwood A, Rafferty H, Moffitt A, Tsitsopoulou A, Gaur S, Holmes T, Backx M. A National Strategy to Diagnose Coronavirus Disease 2019-Associated Invasive Fungal Disease in the Intensive Care Unit. Clin Infect Dis. 2021 Oct 5;73(7):e1634-e1644. doi: 10.1093/cid/ciaa1298. PMID 32860682
- [Derived] Schroeder M, Raboh MA, Nuechtern A, Wichmann D, Stamm J, Hardel T, Rohde H, Christner M, Ozga AK, Steurer S, Jafari C, Klose H, Kluge S, Simon M, Fischer M. Comparison of the Equivalence of Aspergillus Antigen and PCR Results Between Non-Directed Bronchial Lavage and Bronchoalveolar Lavage-A Prospective Exploratory Pilot Study in Critically Ill Patients. Mycoses. 2025 Feb;68(2):e70029. doi: 10.1111/myc.70029. PMID 39900777